CLINICAL TRIAL: NCT03062735
Title: Protocol for a Randomized Controlled Trial Evaluating the Efficacy of Inspiratory Muscle Training on Swimming Performance, Airway Dysfunction and Perceived Breathlessness in Elite Swimmers
Brief Title: Efficacy of Inspiratory Muscle Training on Elite Swimmers
Acronym: PEAK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PEAKNORTE-01-0145-FEDER-000010
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2016-11

CONDITIONS: Reactive Airways Dysfunction Syndrome (Disorder); Muscle Weakness; Dyspnea
MeSH Terms: conditions — Muscle Weakness; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Inspiratory Muscle Training intervention (Sham-IMT) groups during a 3 months training season. A pressure threshold device (POWERbreathe - HaB International Ltd., UK) will be used to IMT. The IMT group will perform 30 inspiratory efforts, 5 times a week, twice daily, for 12 weeks, against a pressure threshold load equivalent to 50% of maximal inspiratory pressure (MIP).
  Interventions: Other: Inspiratory Muscle Training
- Sham Inspiratory Muscle Training (Sham Comparator): Sham-IMT group will follow a similar protocol, except the inspiratory effort that will be made against 15% MIP. The duration of each IMT session will be 30 inspirations. After the initial setting of training loads, the IMT group will be instructed to periodically increase load so that only 30 maneuvers could be completed. The Sham-IMT group will not receive these instructions. All the IMT sessions, in both groups will take place before swimming training and will be supervised throughout the intervention period to ensure that technique and load will be appropriate.
  Interventions: Other: Sham Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — The Inspiratory Muscle Training (IMT) group will perform 30 inspiratory efforts, 5 times a week, twice a day, for 12 weeks, against a pressure threshold load equivalent to 50% of maximal inspiratory pressure.
  Arms: Inspiratory Muscle Training
Other: Sham Inspiratory Muscle Training — The Sham Inspiratory Muscle Training (Sham-IMT) group will perform 30 inspiratory efforts, 5 times a week, twice a day, for 12 weeks, against a pressure threshold load equivalent to 15% of maximal inspiratory pressure.
  Arms: Sham Inspiratory Muscle Training

SUMMARY:
This study is a randomized controlled trial on the efficacy of inspiratory muscle training on swimming performance, airway dysfunction and perceived breathlessness in elite swimmers.

DETAILED DESCRIPTION:
Only a few studies have assessed the impact of Inspiratory Muscle Training (IMT) on swim performance with unclear and inconsistent results. This study aims to evaluate the effect of a 12-week IMT program in swimming performance, airway dysfunction and perceived breathlessness among elite swimmers. Participants will be recruited from the elite competitive Futebol Clube do Porto swimming team. After consent, individuals will be randomly allocated into the IMT or Sham-IMT group. A pressure threshold device will be used to perform the inspiratory training. The IMT group will perform 30 inspiratory efforts, 5 times a week, twice a day, against a pressure threshold load equivalent to 50% of maximal inspiratory pressure (MIP). Sham-IMT group will follow a similar protocol, except for the inspiratory effort that will be made against 15% of MIP. Measures of lung function, swimming performance, airway dysfunction, inspiratory muscle strength and perceived breathlessness will be assessed at the beginning and then in 4 weeks intervals until the end of study period. All outcome measures will be assessed by an investigator who will be not involved in the intervention process. Data will be expressed as mean ± standard deviation (SD) and respective 95% confidence interval. The significance level will be 5% (p˂0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy elite swimmers engaged in competitive training for a minimum period of three years;
* Individuals with no disability;
* Individuals aged between 14 and 40 years.

Exclusion Criteria:

* Individuals presenting co-morbidities or physical impairment that affects regular training;
* Smokers;
* Athletes already in a regular respiratory muscle training program
* Individuals with a predicted forced expiratory volume in the first second (FEV1) below 60%.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Swimming time trials performance | twelve weeks
  Changes in time-trial swim performance

CONTACTS AND LOCATIONS:
Overall Officials: André Moreira, MD, PhD, Principal Investigator — Faculty of Medicine of the University of Porto
Locations (1):
- Faculty of Medicine of Porto University, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No